CLINICAL TRIAL: NCT04243928
Title: Role of Kinesiotape Over Dorsi Flexors Muscles on Balance in Children With Spastic Diplegia (Using Biodex Balance System)
Brief Title: Role of Kinesiotape Over Dorsi Flexors Muscles on Balance in Children With Spastic Diplegia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Samar Samy Ibrahim Hegazy, ROLE OF KINESIOTAPE OVER DORSI FLEXORS MUSCLES ON BALANCE IN CHILDREN WITH SPASTIC DIPLEGIA, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: peadiatrics 123
Record Dates: First submitted 2020-01-22; First posted 2020-01-28 (Actual); Last update posted 2020-01-28 (Actual); Status verified 2017-12

CONDITIONS: Cerebral Palsy
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Intervention Model Description: children rranged from 4 years uo to 10 years with Spastic diplegia
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (Active Comparator): 15 diplegic children received regular exercise program including balance exercise
  Interventions: Other: kinesio taping
- study group (Experimental): 15 diplegic children recieved regular exercise program plus putting kinesiotape
  Interventions: Other: kinesio taping

INTERVENTIONS:
Other: kinesio taping — apply kinesio taping on dorsi flexors muscles

SUMMARY:
To detect the effect of kinesio -tape on balance in children with spastic diplegia.

DETAILED DESCRIPTION:
The use of Kinesio Taping might influence the cutaneous receptors of the sensory motor system, resulting in the improvement of voluntary control and coordination in a physiotherapy program for children with CP. (Yasukawa et al., 2006).

The study will be conducted To investigate the effect of kinesiotape applied on dorsi fexors muscles on improving balance in spastic diplegic children .

ELIGIBILITY:
Inclusion Criteria:

* • Thirty children with spastic diplegia of both genders participated in this study.

  * Theywere selected from the out-patient clinic, faculty of physical therapy, Cairo University.
  * Children height not less than 1 meter to be able to see the screen of the biodex balance system.
  * Their agehad ranged from 4 to 8 years.
  * All patients have mild spasticity according to modified Aschwar scale grade 1 &1+ (Alhusaini, 2010) presented in (Appendix I).
  * All patients wereable to stand alone GMFM presented in (Appendix II).
  * They could understand and follow instructions.
  * All Children used Ankle Foot Orthosis.

Exclusion Criteria:

* • Children with visual or auditory problems.

  * Children with positive sensitivity to kinesiotape.
  * Children with irrivisable muscle contracture at the calf muscles.

Ages: 4 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2019-02-10 (Actual); Primary Completion 2019-08-11 (Actual); Study Completion 2019-10-13 (Actual)

PRIMARY OUTCOMES:
effect of K-Tape on balance | three months
  effect of using K-Tape on dorsi flexors to see its effect on balance

CONTACTS AND LOCATIONS:
Overall Officials: I, Principal Investigator — Cairo University
Locations (1):
- Cairo Univeristy, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No